CLINICAL TRIAL: NCT05276804
Title: The POUR Study: Effects of Neuromuscular Reversal Agents on Postoperative Urinary Retention (POUR) Following Laparoscopic Inguinal Hernia Repair
Brief Title: The POUR (Postoperative Urinary Retention) Study
Acronym: POUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00083113; 01-22-45E (Other: Atrium)
Record Dates: First submitted 2022-03-01; First posted 2022-03-11 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Urinary Retention
Keywords: Sugammadex
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Experimental): Prospective cohort of patients undergoing laparoscopic inguinal hernia repair will receive Sugammadex. Sugammadex will be used for reversal of their neuromuscular blockade. The dosing for Sugammadex is 4mg/kg for a deep reversal and a 2mg/kg for a standard reversal, which will be more common for this study. Sugammadex comes in 200mg/2mL and 500mg/5mL vials. Because of the variability in weight of the patients and the type of reversal needed (deep vs standard), 140 5mL vials will be required.
  Interventions: Drug: Sugammadex
- Retrospective cohort (No Intervention): Retrospective cohort of patients who did not receive Sugammadex

INTERVENTIONS:
Drug: Sugammadex — The dosing for Sugammadex is 4mg/kg for a deep reversal and a 2mg/kg for a standard reversal, which will be more common for this study. Sugammadex comes in 200mg/2mL and 500mg/5mL vials. Because of the variability in weight of the patients and the type of reversal needed (deep vs standard), 140 5mL vials will be required.
  Arms: Sugammadex

SUMMARY:
The primary aim of this study will be to compare the rate of postoperative urinary retention between patients receiving Sugammadex and those receiving traditional reversal agents

DETAILED DESCRIPTION:
Postoperative urinary retention following laparoscopic inguinal hernia repair occurs in approximately one out of ten patients. The more rapid reversal of neuromuscular blockade with Sugammadex has empirically been associated with low rates of postoperative urinary retention. In this study, patients will receive Sugammadex following laparoscopic inguinal hernia repair and then be retrospectively matched against a group of patients who did not receive Sugammadex. The primary aim of this study will be to compare the rate of postoperative urinary retention between patients receiving Sugammadex and those receiving traditional reversal agents (e.g. neostigmine which has a retention rate of 5-11%). We will also examine difference in cost and quality of life between the two groups. Our hypothesis is that the use of Sugammadex will decrease rate of postoperative urinary retention, decrease associated cost, such as need for admission, and not negatively impact quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Undergoing laparoscopic inguinal hernia repair at Carolinas Medical Center by attending surgeons within the Division of Gastrointestinal and Minimally Invasive Surgery
* Unilateral or bilateral inguinal hernia repair; may have concurrent umbilical hernia repair performed
* Agreeable to participation in the study

Exclusion Criteria:

* Patients who are having concurrent ventral or flank hernias repaired at time of operation or are having an inguinal hernia repair along with another operation (e.g.

laparoscopic cholecystectomy)

* End-stage renal disease (Creatinine clearance less than 30)
* Neuromuscular disease
* Prior adverse reactions to Sugammadex
* Patients who do not provide consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant T Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 prospectively enrolled into Sugammadex group 74 retrospectively matched from baseline (non-Sugammadex) group
Period: Overall Study
Arm/Group | Sugammadex | Retrospective Cohort
Started | 97 | 74
Completed | 74 | 74
Not Completed | 23 | 0
Not completed — screen failure | 23 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Retrospective Cohort | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at time of surgery, in years
  Years | 59.4 (15.5) | 59.2 (14.6) | 59.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Count and percentage of males and females
  Participants
    Female | 5 | 4 | 9
    Male | 69 | 70 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 11 | 12 | 23
    White | 62 | 59 | 121
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 3 | 4
History of BPH (Benign prostatic hyperplasia) [Count of Participants; unit: Participants] — Count of BPH history
  Participants
    Yes | 10 | 15 | 25
    No | 64 | 59 | 123
Side of Inguinal Repair [Count of Participants; unit: Participants] — Bilateral vs Unilateral Repair
  Participants
    Unilateral | 44 | 47 | 91
    Bilateral | 30 | 27 | 57
Surgical Repair Technique [Count of Participants; unit: Participants] — Planned operative technique for inguinal hernia repair
  Participants
    Laparoscopic | 35 | 59 | 94
    Robotic | 39 | 15 | 54
Tobacco Status [Count of Participants; unit: Participants] — Tobacco status of the participant at time baseline
  Participants
    Never | 39 | 42 | 81
    Former | 30 | 21 | 51
    Current | 5 | 11 | 16
Primary vs Recurrent Repair [Count of Participants; unit: Participants] — Primary or recurrent hernia repair
  Participants
    Primary | 63 | 64 | 127
    Recurrent | 11 | 10 | 21
Diabetes Status [Count of Participants; unit: Participants] — Diabetes Status at time of surgery
  Participants
    Yes | 6 | 1 | 7
    No | 68 | 73 | 141
Steroids Use [Count of Participants; unit: Participants] — Steroids use at time of surgery
  Participants
    Yes | 5 | 8 | 13
    No | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urinary Retention
Description: Urinary retention is defined as the inability to void at six hours postoperatively, which will be recorded in the postoperative recovery area and the same definition for urinary retention will be applied to the comparative retrospective cohort
Time Frame: 6 hours postop
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
Participants
  Yes | 0 | 11
  No | 74 | 63

2. Secondary Outcome: Length of Stay (Days)
Description: Patients will be followed from post surgery until discharge to determine the interim time
Time Frame: From post op to discharge (up to 365 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
Days | 0.0 (0.1) | 0.3 (0.9)

3. Secondary Outcome: Hospital Cost
Description: Patient costs associated with procedure and hospital stay
Time Frame: At discharge (up to 365 days)
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
USD | 57954 (13448) | 54970 (19324)

4. Other Pre Specified Outcome: Quality of Life Survey
Description: Quality of life survey given post hernia repair to evaluate mesh sensation, pain and movement limitations. 23 total items. Each item is scored 0 (no symptoms) to 5 (disabling symptoms). Total score range is 0-115 with a low score indicating surgery had no negative impact on quality of life.
Time Frame: Week 2
Population: This outcome measure type was entered incorrectly when the study was initially registered. The QOL survey should have been designated as "other."
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Operation Time
Description: Number of minutes the operation lasted
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
minutes | 105.9 (26.8) | 102.1 (51.3)

6. Other Pre Specified Outcome: Morphine Milligram Equivalents
Description: Morphine milligram equivalents (MME) represents the potency of an opioid dose relative to morphine. MME is intended to help clinicians make safe, appropriate decisions concerning changes to opioid regimens.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
milligrams | 38.3 (11.9) | 38.0 (17.8)

7. Other Pre Specified Outcome: Number of Participants With Clean Wounds at Follow Up
Description: Number of participants with clean wounds based on the Center for Disease Control and Prevention (CDC) Wound guidelines. CDC wound classification options are Clean, Clean-Contaminated, Contaminated, and Dirty/Infected.
Time Frame: Up to Week 2
Measure: Number; unit: participants
Arm/Group | Sugammadex | Retrospective Cohort
Number analyzed (Participants) | 74 | 74
participants | 74 | 74

ADVERSE EVENTS:
Time Frame: Up to Week 2
Description: Number of adverse events reported
Arm/Group | Sugammadex | Retrospective Cohort
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT05276804/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT05276804/ICF_002.pdf